CLINICAL TRIAL: NCT01789398
Title: Double Blind Randomized Study to Assess the Efficacy of BF2.649 Compared to Placebo in add-on to Sodium Oxybate in the Treatment of Narcoleptic Patients With Residual Excessive Daytime Sleepiness (EDS) During 8 Weeks
Brief Title: Patient Narcoleptic Treated With BF2.649 (Pitolisant) in add-on to Sodium Oxybate (HARMONY IV)
Acronym: HARMONY IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P10-01 / BF2.649; 2011-000084-27 (EudraCT Number)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF2.649 (pitolisant) (Experimental): BF2.649 (5mg, 10mg, 20mg or 40mg) in capsules
  Interventions: Drug: BF2.649
- placebo (Placebo Comparator): Placebo of BF2.649 (5mg, 10mg, 20mg or 40mg) in capsules
  Interventions: Drug: BF2.649

INTERVENTIONS:
Drug: BF2.649 — BF2.649 is provided in capsules. Patients should take 1 capsules per day with a glass of water. They will be instructed to take 1 capsule in the morning (after waking up, before breakfast).
  Other Names: pitolisant

SUMMARY:
This is a multicentric international phase III, double blind randomized study assessing efficacy and safety in parallel group of BF2.649 (pitolisant) compared to placebo in add-on to sodium oxybate of narcoleptic patients with residual Excessive Daytime Sleepiness (EDS) during 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18 years old and over.
* Patients with a diagnosis of narcolepsy according to the International Classification of Sleep Disorders (ICSD-2) criteria
* Patients treated with sodium oxybate (Xyrem®) with a stable dosage for at least 2 months prior to the trial.
* Patients complaining of residual EDS
* Patient should be free of non authorized drugs or discontinue any psychostimulant medication at least 3 weeks before randomization (V2).
* Females of child-bearing potential must use a medically accepted effective method of birth control, agree to continue this method for the duration of the study and be negative to serum pregnancy test performed at the screening visit. Females should not be breast-feeding patient.
* In the opinion of the investigator, the patient must have adequate support to comply with the entire study requirements as described in the protocol (e.g. transportation to and from trial site, self rating scales, drug compliance, scheduled visits, etc).
* Patient must have voluntarily expressed a willingness to participate in this study, signed and dated an informed consent prior to beginning this protocol required procedures.

Exclusion Criteria:

* Psychiatric and neurological disorders, other than narcolepsy/cataplexy, such as moderate or severe psychosis or dementia, bipolar illness, severe anxiety, clinical severe depression (BDI ≥ 16) with suicidal risk (item G BDI > 0), or depression treated for less than 8 weeks, history of seizure disorder or other problem that in the investigator's opinion would preclude the patient's participation and completion of this trial or comprise reliable representation of subjective symptoms.
* Patients working in an occupation requiring variable shift work or routine night shifts.
* Patients with an untreated sleep apnea disorder (defined as an apnea index > 10/h or an apnea/hypopnea index>15/h) or who have any other cause of daytime sleepiness.
* Use of hypnotics, tranquilizers, sedating antihistamines, psychostimulants for the treatment of EDS (amphetamine and amphetamine-like CNS stimulants, modafinil, methylphenidate or others), benzodiazepines, anticonvulsants or clonidine will not be accepted at least 3 weeks before randomization (V2) and during study.
* Current or recent (within one year) history of a substance abuse or dependence disorder including alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
* Other active clinically significant illness, including unstable cardiovascular, or neoplasic pathology which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise the study participation.
* Patient with a known history of long QTc syndrome (e.g. syncope or arythmia) or presenting any significant serious abnormality of the ECG (e.g. recent myocardial infarction), or QTc interval strictly higher than 450 ms (electrocardiogram Bazett's corrected).
* Patients with Severe Hepatic Impairment or with Severe Renal Impairment, or with any other significant abnormality in the physical examination or clinical laboratory results.
* Known hypersensitivity to the tested treatment including active substance and excipients.
* Patients participating in an other study and the use of any investigational therapy within the 30 days prior to the entry in this study.
* Patient without any medical care insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Efficacy on EDS as measured by ESS ( Epworth Sleepiness Scale) | 8 weeks
  based on the ESS score change from baseline to final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, Study Chair — Hôpital Gui de Chauliac - 80, avenue A. Fliche , 34295 Montpellier cedex 5 - FRANCE
Locations (1):
- CHU Montpellier, Montpellier, Montpellier, France